CLINICAL TRIAL: NCT00430508
Title: Efficacy and Safety of Hydrochlorothiazide (HCTZ) Used as Add-on Therapy in Moderately to Severely Hypertensive Patients Not Adequately Controlled by Olmesartan Medoxomil (OM) 40 mg Monotherapy
Brief Title: Use of the Combination of Olmesartan and Hydrochlorothiazide in Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Bettina Ammentorp, Daichi Sankyo Europe, GmbH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS866CM-B-E301
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Results first posted 2009-06-17 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2009-06

CONDITIONS: Essential Hypertension
Keywords: Moderate-to-Severe Hypertension; Essential Hypertension; Combination Therapy; Fixed-Combination Dose
MeSH Terms: conditions — Essential Hypertension | interventions — Olmesartan Medoxomil; Hydrochlorothiazide; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 4 (Experimental): olmesartan medoxomil (OM) /hydrochlorothiazide (HCTZ) Tablet 40mg/0mg + 20mg/12.5mg matching placebo tablet once daily for 8 weeks
  Interventions: Drug: olmesartan medoxomil (OM)/hydrochlorothiazide (HCTZ) tablets and placebo
- 1 (Experimental): olmesartan medoxomil (OM) /hydrochlorothiazide (HCTZ) tablets 40mg/25mg + 20mg/12.5mg matching placebo tablet once daily for 8 weeks
  Interventions: Drug: olmesartan medoxomil/hydrochlorothiazide tablets
- 3 (Experimental): olmesartan medoxomil (OM)/hydrochlorothiazide (HCTZ) tablets 20mg/12.5mg + 40mg/0mg matching placebo tablet once daily for 8 weeks
  Interventions: Drug: olmesartan medoxomil/hydrochlorothiazide tablets
- 2 (Experimental): olmesartan medoxomil (OM)/hydrochlorothiazide (HCTZ) tablets 40mg/12.5mg + 20mg/12.5mg matching placebo tablet once daily for 8 weeks
  Interventions: Drug: olmesartan medoxomil (OM)/hydrochlorothiazide (HCTZ) tablets

INTERVENTIONS:
Drug: olmesartan medoxomil (OM)/hydrochlorothiazide (HCTZ) tablets and placebo — olmesartan medoxomil (OM)/hydrochlorothiazide (HCTZ) Tablet 40mg/0mg + 20mg/12.5mg matching placebo tablet once daily for 8 week
  Arms: 4
Drug: olmesartan medoxomil (OM)/hydrochlorothiazide (HCTZ) tablets — olmesartan medoxomil (OM)/hydrochlorothiazide (HCTZ) tablets 40mg/12.5mg + 20mg/12.5mg matching placebo tablet once daily for 8 weeks
  Arms: 2
Drug: olmesartan medoxomil/hydrochlorothiazide tablets — olmesartan medoxomil (OM)/hydrochlorothiazide (HCTZ) tablets 40mg/25mg + 20mg/12.5mg matching placebo tablet once daily for 8 weeks
  Arms: 1
Drug: olmesartan medoxomil/hydrochlorothiazide tablets — olmesartan medoxomil (OM)/hydrochlorothiazide (HCTZ) tablets 20mg/12.5mg + 40mg/0mg matching placebo tablet once daily for 8 weeks
  Arms: 3

SUMMARY:
The study will evaluate the blood pressure lowering effects of two different dosages of the combination of olmesartan and hydrochlorothiazide in patients with moderate or severe high blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Europeans aged 18 years or older with moderate to severe hypertension (HTN)

Exclusion Criteria:

* Female patients of childbearing potential pregnant, lactating or planning to become pregnant during the trial period.
* Patients with serious disorders which may limit the ability to evaluate the efficacy or safety of the study medication, including cerebrovascular, cardiovascular, renal, respiratory, hepatic, gastrointestinal, endocrine or metabolic, haematological or oncological, neurological and psychiatric diseases.
* Patients having a history of the following within the last six months:

  * myocardial infarction,
  * unstable angina pectoris,
  * percutaneous coronary intervention,
  * severe heart failure,
  * hypertensive encephalopathy,
  * cerebrovascular accident (stroke) or
  * transient ischaemic attack.
* Patients with clinically significant abnormal laboratory values at screening.
* Patients with secondary HTN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 972 (Actual)
Dates: Start 2007-02; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor Lars Christian Rump, M.D., Study Chair — University of Ruhr-Bochum
Locations (55):
- Bulgaria (2):
  - Pleven
  - Sofia
- Czechia (14):
  - Beroun
  - Brno
  - Chrudim
  - Hradec Králové
  - Jindřichův Hradec
  - Kutná Hora
  - Ostrava
  - Pardubice
  - Pilsen
  - Prague
  - Příbram
  - Řevnice
  - Sokolov
  - Trutnov
- France (3):
  - Langres
  - Paris
  - Pessac
- Germany (11):
  - Berlin
  - Bochum
  - Dietzenbach
  - Franfurt
  - Friedberg
  - Ingelheim
  - Karlsbad
  - Leipzig
  - Offenbach
  - Siegen
  - Stuhr-Brinkum
- Poland (12):
  - Elblag
  - Gdansk
  - Inowrocław
  - Katowice
  - Krakow
  - Linia
  - Lodz
  - Oława
  - Poznan
  - Warsaw
  - Wroclaw
  - Zamość
- Spain (4):
  - Girona
  - Granada
  - Madrid
  - Oviedo
- Ukraine (9):
  - Dnipro
  - Donetsk
  - Kharkiv
  - Kiev
  - Lviv
  - Odesa
  - Uzhhorod
  - Vinnytsia
  - Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Rosenbaum D, Girerd X. Olmesartan medoxomil combined with hydrochlorothiazide improves 24-hour blood pressure control in moderate-to-severe hypertension. Curr Med Res Opin. 2012 Feb;28(2):179-86. doi: 10.1185/03007995.2011.644626. Epub 2012 Jan 9. PMID 22114906

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 78 investigative sites screened patients in Europe (19 in Czech Republic, 11 in Germany, 8 in Bulgaria, 5 in Spain, 20 in Ukraine, 1 in France and 14 in Poland).
  Sites were either hospitals or general practitioners. First patient in: 17 January 2007 Last patient out: 30 March 2008
Pre-assignment Details: Trial is 2-week taper-off phase and 2 treatment periods. Period I-8-week open-label, OM 40mg. End of Period I, only non-responders randomised to Period II. Blood Pressure controlled patients discontinued. Period II-8-week double-blind four randomized treatment arms. Participant flow is Period II. 972 completed period I, 971 started period II.
Groups:
- OM/HCTZ 40/25mg + 20/12.5 Matching Placebo: olmesartan medoxomil/Hydrochlorothizaide 40/25mg tablets, once daily for 8 weeks
- OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo: olmesartan medoxomil/Hydrochlorothizaide 40/12.5mg tablets, once daily for 8 weeks
- OM/HCTZ 20/12.5mg + 40/0 Matching Placebo: olmesartan medoxomil/Hydrochlorothizaide 20/12.5mg tablets, once daily for 8 weeks
- OM/HCTZ 40/0mg + 20/12.5 Matching Placebo: olmesartan medoxomil/Hydrochlorothizaide 40/0mg tablets, once daily for 8 weeks
Period: Overall Study
Arm/Group | OM/HCTZ 40/25mg + 20/12.5 Matching Placebo | OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo | OM/HCTZ 20/12.5mg + 40/0 Matching Placebo | OM/HCTZ 40/0mg + 20/12.5 Matching Placebo
Started | 140 | 278 | 279 | 274
Completed | 137 | 272 | 266 | 269
Not Completed | 3 | 6 | 13 | 5
Not completed — Adverse Event | 2 | 3 | 5 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1
Not completed — responder at visit 4 | 0 | 0 | 2 | 0
Not completed — conmed-BP-pulse-ABPM withdrawal criteria | 0 | 1 | 2 | 1
Not completed — Other | 1 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OM/HCTZ 40/25mg + 20/12.5 Matching Placebo | OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo | OM/HCTZ 20/12.5mg + 40/0 Matching Placebo | OM/HCTZ 40/0mg + 20/12.5 Matching Placebo | Total
Number analyzed (Participants) | 140 | 278 | 279 | 274 | 971
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 122 | 240 | 233 | 238 | 833
  >=65 years | 18 | 38 | 46 | 36 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (8.17) | 53.7 (9.77) | 55.2 (9.47) | 54.1 (8.92) | 54.5 (9.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 105 | 100 | 115 | 372
  Male | 88 | 173 | 179 | 159 | 599
Race/Ethnicity, Customized [Number; unit: participants]
  European | 140 | 278 | 278 | 274 | 970.0
  Other | 0 | 0 | 1 | 0 | 1.0

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Trough Sitting Diastolic Blood Pressure From Week 8(Baseline) to Week 16
Description: Change = Week 16 - Week 8 (baseline).
Time Frame: 8 weeks, change = week 16 - week 8
Population: Full Analysis Set-Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- OM/HCTZ 40/25mg + 20/12.5 Matching Placebo: olmesartan medoxomil/HCTZ Tablet 40mg/25mg + 20mg/12.5mg matching placebo tablet once daily for 8 weeks
- OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo: olmesartan medoxomil/hydrochlorothiazide tablets 40mg/12.5mg + 20mg/12.5mg matching placebo tablet once daily for 8 weeks
- OM/HCTZ 20/12.5mg + 40/0 Matching Placebo: olmesartan medoxomil/hydrochlorothiazide tablets 20mg/12.5mg + 40mg/0mg matching placebo tablet once daily for 8 weeks
- OM/HCTZ 40/0mg + 20/12.5 Matching Placebo: olmesartan medoxomil/hydrochlorothiazide tablets 40mg/0mg + 20mg/12.5mg matching placebo tablet once daily for 8 weeks
Arm/Group | OM/HCTZ 40/25mg + 20/12.5 Matching Placebo | OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo | OM/HCTZ 20/12.5mg + 40/0 Matching Placebo | OM/HCTZ 40/0mg + 20/12.5 Matching Placebo
Number analyzed (Participants) | 140 | 277 | 279 | 274
mm Hg | -11.16 (8.796) | -9.13 (8.622) | -8.10 (7.968) | -5.66 (8.546)
Statistical Analysis 1: Comparison: OM/HCTZ 40/25mg + 20/12.5 Matching Placebo vs OM/HCTZ 40/0mg + 20/12.5 Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -5.3, 95% CI [-6.97 to -3.6]
Statistical Analysis 2: Comparison: OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo vs OM/HCTZ 40/0mg + 20/12.5 Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -3.4, 95% CI [-4.79 to -2.03]
Statistical Analysis 3: Comparison: OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo vs OM/HCTZ 20/12.5mg + 40/0 Matching Placebo; Test type: Superiority or Other; p = 0.1788, ANCOVA; Mean Difference (Net) = -0.9, 95% CI [-2.32 to 0.43]

2. Secondary Outcome: Change in Mean Trough Sitting Diastolic Blood Pressure From Week 8(Baseline) to Week 12.
Description: Change = Week 12 - Week 8 (baseline).
Time Frame: 4 weeks, change = week 12 - week 8
Population: Full Analysis Set-Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | OM/HCTZ 40/25mg + 20/12.5 Matching Placebo | OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo | OM/HCTZ 20/12.5mg + 40/0 Matching Placebo | OM/HCTZ 40/0mg + 20/12.5 Matching Placebo
Number analyzed (Participants) | 140 | 277 | 279 | 274
mm Hg | -8.74 (7.879) | -7.72 (7.606) | -6.66 (7.090) | -4.47 (7.197)
Statistical Analysis 1: Comparison: OM/HCTZ 40/25mg + 20/12.5 Matching Placebo vs OM/HCTZ 40/0mg + 20/12.5 Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -4.1, 95% CI [-5.54 to -2.6]
Statistical Analysis 2: Comparison: OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo vs OM/HCTZ 40/0mg + 20/12.5 Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -3.2, 95% CI [-4.39 to -1.98]
Statistical Analysis 3: Comparison: OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo vs OM/HCTZ 20/12.5mg + 40/0 Matching Placebo; Test type: Superiority or Other; p = 0.1081, ANCOVA; Mean Difference (Net) = -1.0, 95% CI [-2.19 to 0.22]

3. Secondary Outcome: Change in Mean Trough Sitting Systolic Blood Pressure From Week 8(Baseline) to Week 16.
Description: Change = Week 16 - Week 8 (baseline).
Time Frame: 8 weeks, change = week 16 - week 8
Population: Full Analysis Set-Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | OM/HCTZ 40/25mg + 20/12.5 Matching Placebo | OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo | OM/HCTZ 20/12.5mg + 40/0 Matching Placebo | OM/HCTZ 40/0mg + 20/12.5 Matching Placebo
Number analyzed (Participants) | 140 | 277 | 279 | 274
mm Hg | -16.17 (13.444) | -13.52 (14.533) | -11.46 (13.673) | -8.85 (13.537)
Statistical Analysis 1: Comparison: OM/HCTZ 40/25mg + 20/12.5 Matching Placebo vs OM/HCTZ 40/0mg + 20/12.5 Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -7.4, 95% CI [-10.13 to -4.66]
Statistical Analysis 2: Comparison: OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo vs OM/HCTZ 40/0mg + 20/12.5 Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -5.2, 95% CI [-7.4 to -2.91]
Statistical Analysis 3: Comparison: OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo vs OM/HCTZ 20/12.5mg + 40/0 Matching Placebo; Test type: Superiority or Other; p = 0.0255, ANCOVA; Mean Difference (Net) = -2.6, 95% CI [-4.79 to -0.31]

4. Secondary Outcome: Change in Mean Trough Sitting Systolic Blood Pressure From Week 8(Baseline) to Week 12.
Description: Change = Week 12 - Week 8 (baseline).
Time Frame: 4 weeks, change = week 12 - week 8
Population: Full Analysis Set-Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | OM/HCTZ 40/25mg + 20/12.5 Matching Placebo | OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo | OM/HCTZ 20/12.5mg + 40/0 Matching Placebo | OM/HCTZ 40/0mg + 20/12.5 Matching Placebo
Number analyzed (Participants) | 140 | 277 | 279 | 274
mm Hg | -13.16 (13.337) | -10.90 (12.297) | -9.65 (11.743) | -6.60 (10.932)
Statistical Analysis 1: Comparison: OM/HCTZ 40/25mg + 20/12.5 Matching Placebo vs OM/HCTZ 40/0mg + 20/12.5 Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -6.6, 95% CI [-9.00 to -4.26]
Statistical Analysis 2: Comparison: OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo vs OM/HCTZ 40/0mg + 20/12.5 Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -4.8, 95% CI [-6.70 to -2.81]
Statistical Analysis 3: Comparison: OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo vs OM/HCTZ 20/12.5mg + 40/0 Matching Placebo; Test type: Superiority or Other; p = 0.0812, ANCOVA; Mean Difference (Net) = -1.7, 95% CI [-3.66 to 0.21]

5. Secondary Outcome: Number of Patients Achieving Target Blood Pressure at Week 16
Description: Target Blood Pressure is diastolic blood pressure (dBP) < 90 mmHg and systolic blood pressure (sBP) < 140 mmHg for non-diabetics, and dBP < 80 mmHg and sBP < 130 mmHg for diabetics
Time Frame: 8 weeks
Population: Full Analysis Set-Last Observation Carried Forward
Measure: Number; unit: participants
Arm/Group | OM/HCTZ 40/25mg + 20/12.5 Matching Placebo | OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo | OM/HCTZ 20/12.5mg + 40/0 Matching Placebo | OM/HCTZ 40/0mg + 20/12.5 Matching Placebo
Number analyzed (Participants) | 140 | 277 | 279 | 274
participants | 59 | 110 | 88 | 68
Statistical Analysis 1: Comparison: OM/HCTZ 40/25mg + 20/12.5 Matching Placebo vs OM/HCTZ 40/0mg + 20/12.5 Matching Placebo; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 2.67, 95% CI [1.69 to 4.21]
Statistical Analysis 2: Comparison: OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo vs OM/HCTZ 40/0mg + 20/12.5 Matching Placebo; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 2.20, 95% CI [1.50 to 3.24]
Statistical Analysis 3: Comparison: OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo vs OM/HCTZ 20/12.5mg + 40/0 Matching Placebo; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 1.55, 95% CI [1.07 to 2.25]

6. Secondary Outcome: Change in Mean 24-hour Ambulatory Blood Pressure Monitoring Diastolic Blood Pressure From Week 8(Baseline) to Week 16.
Description: Change = Week 16 - Week 8 (baseline).
Time Frame: 8 weeks, change = week 16 - week 8
Population: Full Analysis Set-Observed Cases
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | OM/HCTZ 40/25mg + 20/12.5 Matching Placebo | OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo | OM/HCTZ 20/12.5mg + 40/0 Matching Placebo | OM/HCTZ 40/0mg + 20/12.5 Matching Placebo
Number analyzed (Participants) | 120 | 250 | 241 | 249
mm Hg | -7.2 (7.62) | -5.3 (8.60) | -4.1 (9.07) | -2.0 (7.64)
Statistical Analysis 1: Comparison: OM/HCTZ 40/25mg + 20/12.5 Matching Placebo vs OM/HCTZ 40/0mg + 20/12.5 Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -5.1, 95% CI [-6.78 to -3.36]
Statistical Analysis 2: Comparison: OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo vs OM/HCTZ 40/0mg + 20/12.5 Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -3.2, 95% CI [-4.54 to -1.78]
Statistical Analysis 3: Comparison: OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo vs OM/HCTZ 20/12.5mg + 40/0 Matching Placebo; Test type: Superiority or Other; p = 0.1452, ANCOVA; Mean Difference (Net) = -1.0, 95% CI [-2.43 to 0.36]

7. Secondary Outcome: Change in Mean Daytime Ambulatory Blood Pressure Monitoring Diastolic Blood Pressure From Week 8(Baseline) to Week 16.
Description: Change = Week 16 - Week 8 (baseline).
Time Frame: 8 weeks, change = week 16 - week 8
Population: Full Analysis Set-Observed Cases
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | OM/HCTZ 40/25mg + 20/12.5 Matching Placebo | OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo | OM/HCTZ 20/12.5mg + 40/0 Matching Placebo | OM/HCTZ 40/0mg + 20/12.5 Matching Placebo
Number analyzed (Participants) | 120 | 250 | 241 | 249
mm Hg | -7.0 (8.06) | -5.5 (9.10) | -4.0 (9.34) | -1.8 (8.39)
Statistical Analysis 1: Comparison: OM/HCTZ 40/25mg + 20/12.5 Matching Placebo vs OM/HCTZ 40/0mg + 20/12.5 Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -5.0, 95% CI [-6.79 to -3.17]
Statistical Analysis 2: Comparison: OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo vs OM/HCTZ 40/0mg + 20/12.5 Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -3.3, 95% CI [-4.79 to -1.87]
Statistical Analysis 3: Comparison: OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo vs OM/HCTZ 20/12.5mg + 40/0 Matching Placebo; Test type: Superiority or Other; p = 0.1629, ANCOVA; Mean Difference (Net) = -1.0, 95% CI [-2.52 to 0.42]

8. Secondary Outcome: Change in Mean Night-time Ambulatory Blood Pressure Monitoring Diastolic Blood Pressure From Week 8(Baseline) to Week 16.
Description: Change = Week 16 - Week 8 (baseline).
Time Frame: 8 weeks, change = week 16 - week 8
Population: Full Analysis Set-Observed Cases
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | OM/HCTZ 40/25mg + 20/12.5 Matching Placebo | OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo | OM/HCTZ 20/12.5mg + 40/0 Matching Placebo | OM/HCTZ 40/0mg + 20/12.5 Matching Placebo
Number analyzed (Participants) | 120 | 250 | 241 | 249
mm Hg | -7.9 (9.51) | -4.5 (9.90) | -4.2 (10.61) | -2.3 (8.47)
Statistical Analysis 1: Comparison: OM/HCTZ 40/25mg + 20/12.5 Matching Placebo vs OM/HCTZ 40/0mg + 20/12.5 Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -5.5, 95% CI [-7.40 to -3.62]
Statistical Analysis 2: Comparison: OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo vs OM/HCTZ 40/0mg + 20/12.5 Matching Placebo; Test type: Superiority or Other; p < 0.0009, ANCOVA; Mean Difference (Net) = -2.6, 95% CI [-4.12 to -1.07]
Statistical Analysis 3: Comparison: OM/HCTZ 40/12.5mg + 20/12.5 Matching Placebo vs OM/HCTZ 20/12.5mg + 40/0 Matching Placebo; Test type: Superiority or Other; p = 0.1985, ANCOVA; Mean Difference (Net) = -1.0, 95% CI [-2.55 to 0.53]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results of Study shall not be published without prior express written consent and approval of Sponsor. If Contractor wishes to use data generated at Sites by Investigator, such data includes but not limited to data used in collection of metrics, copy of any intended publication, details of use must be sent in writing to Quintiles and Sponsor for review. Sponsor has right to change proposed publication and/or prohibit publication and Contractor must comply with requirements of Sponsor